CLINICAL TRIAL: NCT05383261
Title: The Impact of the Social Factors and Medical Rehabilitation Program to Address the Implications on Kidney Failure Disease in Hail Region (Under the Vision 2030)
Brief Title: The Impact of the Social Factors and Rehabilitation Program to Address the Implications on Kidney Failure in Hail
Status: Completed | Type: Observational
Sponsor: University of Hail (Other)
Responsible Party: Principal Investigator, Ahmed Abdelmoniem Ibrahim, aassoci prof, University of Hail
Other Study IDs: RG-191348
Record Dates: First submitted 2022-05-16; First posted 2022-05-20 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Chronic Renal Disease
Keywords: Renal failure patients -Saudi community - social program
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- control: patients will take medical treatment only
  patients will receive medical treatment in addition to aerobic exercises
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — aerobic and resisted ex

SUMMARY:
The aims of our study to evaluate the effect of social factors and medical rehabilitation program on kidney function and quality of life among chronic kidney disease patients.

DETAILED DESCRIPTION:
1. This study aims to evaluate the effect of social factors and medical rehabilitation program on kidney function and quality of life among chronic kidney disease patients.
2. Identify the health problems facing patients with kidney failure in Hail region.
3. Detect the reality of the problems facing patients with kidney failure in Hail region and ways to reduce them.
4. Identify the family, psychological, economic and social problems facing patients with kidney failure in Hail region.

ELIGIBILITY:
Inclusion Criteria:

participants with CKD stages (3 and 4) will be participated in this study, their ages ranged from 40 to 60 years. Both sexes will be included.

Participants should be: Saudi persons living in Hail City, married, both genders,

Exclusion Criteria:

* (1) Severe chronic cardiac problems. (2) Chronic chest disease. (3) Chronic inflammatory orthopedic disorders and rheumatoid arthritis. (4) Mental impairments.

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: participants with CKD stages (3 and 4) will be participated in this study, their ages ranged from 40 to 60 years. Both sexes will be included.
  Participants should be: Saudi persons living in Hail City, married, both genders,
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
6-minute walk test (6MWT). And Kidney Disease and Quality of Life (KDQOL™-36) | after 6 week
  6-minute walk test (6MWT). And Kidney Disease and Quality of Life (KDQOL™-36)

SECONDARY OUTCOMES:
muscle power of lower limb | after 6 week
  functional muscle test

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hail, Hail, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: hhhhhh — https://pubmed.ncbi.nlm.nih.gov/19240646/
- See also: hhhhh — https://pubmed.ncbi.nlm.nih.gov/15526912/